CLINICAL TRIAL: NCT02314403
Title: Renal Allograft Tolerance Through Mixed Chimerism (Belatacept)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Tatsuo Kawai, MD, PhD, Associate Professor of Surgery, Harvard Medical School, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGH Tolerance Trial
Record Dates: First submitted 2014-12-05; First posted 2014-12-11 (Estimated); Results first posted 2021-09-02 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Kidney Failure, Chronic; Renal Insufficiency
Keywords: ESRD
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency | interventions — Abatacept; Rituximab; Whole-Body Irradiation; Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combined Bone Marrow and Kidney Transplantation (Experimental): Recipients will receive a conditioning regimen that starts with Rituximab on day -7 (and days -2, 5, 12), Whole Body Irradiation 1.5 Gy x2 on study days -6 and -5, followed by ATG on Days -2, -1, 0. Belatacept 10mg/kg on Days 0, 3, 10, 17, 24, 38, 52. Thymic irradiation (7 Gy) will be given on study day -1, and combined renal and bone marrow transplant will be done on study day 0. Prednisone will be started at 2 mg/kg on day 4 and tapered off by day 20. Tacrolimus will be administered on study days -1 through 60, and then tapered if weaning criteria are met.
  Interventions: Drug: Belatacept; Drug: ATG; Drug: Rituximab; Radiation: Total Body Irradiation; Radiation: Thymic Irradiation; Procedure: Combined Bone Marrow/Kidney Transplantation

INTERVENTIONS:
Drug: Belatacept — A selective T-cell (lymphocyte) costimulation blocker
Drug: ATG — A T-Cell Depleting Agent
Drug: Rituximab — B-Cell Depleting Agent
Radiation: Total Body Irradiation
Radiation: Thymic Irradiation
Procedure: Combined Bone Marrow/Kidney Transplantation

SUMMARY:
This study will examine the safety and effectiveness of a combination kidney and bone marrow transplant from a haplo-identical related donor. An investigational medication and other treatments will be given prior to and after the transplant to help protect the transplanted kidney from being attacked by the body's immune system

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-60 years of age
* Candidate for a living-donor renal allograft from an HLA mismatched donor
* First or second transplant with either a living donor or cadaveric transplant as the first transplant.
* Use of FDA-approved methods of contraception by all recipients from the time that study treatment begins until 104 weeks (24 months) after renal transplantation.
* Ability to understand and provide informed consent.
* Serologic evidence of prior exposure to EBV.

Exclusion Criteria:

* ABO blood group-incompatible renal allograft.
* Evidence of anti-HLA antibody within 60 days prior to transplant as assessed by routine methodology (AHG and/or ELISA)
* Leukopenia or thrombocytopenia.
* Positive for HIV-1, hepatitis B core antigen, or hepatitis C virus; or positivity for hepatitis B surface antigen.
* Cardiac ejection fraction < 40% or clinical evidence of insufficiency.
* Forced expiratory volume FEV1 < 50% of predicted.
* Lactation or pregnancy.
* History of cancer other than basal cell carcinoma of the skin or carcinoma in situ of the cervix.
* Underlying renal disease etiology with a high risk of disease recurrence in the transplanted kidney (such as focal segmental glomerulosclerosis, type I or II membranoprolifertive glomerulonephritis).
* Prior dose-limiting radiation therapy.
* Known genetic disease or family history that may result in greater sensitivity to the effects of irradiation, or a physical deformity that would preclude adequate shielding or appropriate dosing during the irradiation component of the conditioning regimen.
* Enrollment in other investigational drug studies within 30 days prior to enrollment.
* Abnormal (>2 times lab normal) values for (a) liver function chemistries (ALT, AST, AP), (b) bilirubin, (c) coagulation studies (PT, PTT).
* Allergy or sensitivity to any component of belatacept, ATG, tacrolimus, or rituximab.
* Maintenance immunosuppression within 3 months prior to conditioning other than physiological doses of steroids, defined as ≤ 50 mg of hydrocortisone or dose equivalent.
* The presence of any medical condition that the investigator deems incompatible with participation in the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2015-02; Primary Completion 2021-03 (Actual); Study Completion 2021-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuo Kawai, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Kawai T, Cosimi AB, Sachs DH. Preclinical and clinical studies on the induction of renal allograft tolerance through transient mixed chimerism. Curr Opin Organ Transplant. 2011 Aug;16(4):366-71. — http://www.ncbi.nlm.nih.gov/pubmed/21666482?dopt=Abstract
- See also: Sachs DH, Sykes M, Kawai T, Cosimi AB. Immuno-intervention for the induction of transplantation tolerance through mixed chimerism. Semin Immunol. 2011 Jun;23(3):165-73. — http://www.ncbi.nlm.nih.gov/pubmed/21839648?dopt=Abstract
- See also: Kawai T, (et.al.) HLA-mismatched renal transplantation without maintenance immunosuppression. N Engl J Med. 2008 Jan 24;358(4):353-61. — http://www.ncbi.nlm.nih.gov/pubmed/18216355?dopt=Abstract

RESULTS

PARTICIPANT FLOW:
Groups:
- Combined Bone Marrow and Kidney Transplantation: Recipients will receive a conditioning regimen that starts with Rituximab on day -7 (and days -2, 5, 12), Whole Body Irradiation 1.5 Gy x2 on study days -6 and -5, followed by ATG on Days -2, -1, 0. Belatacept 10mg/kg on Days 0, 3, 10, 17, 24, 38, 52. Thymic irradiation (7 Gy) will be given on study day -1, and combined renal and bone marrow transplant will be done on study day 0. Prednisone will be started at 2 mg/kg on day 4 and tapered off by day 20. Tacrolimus will be administered on study days -1 through 60, and then tapered if weaning criteria are met.
  Belatacept: A selective T-cell (lymphocyte) costimulation blocker
  ATG: A T-Cell Depleting Agent
  Rituximab: B-Cell Depleting Agent
  Total Body Irradiation
  Thymic Irradiation
  Combined Bone Marrow/Kidney Transplantation
Period: Overall Study
Arm/Group | Combined Bone Marrow and Kidney Transplantation
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Combined Bone Marrow and Kidney Transplantation
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Withdrawal of Immunosuppression
Description: The Primary Outcome is: The induction of transient mixed chimerism and renal allograft tolerance (24 consecutive months off of immunosuppression)
Time Frame: 5 Years
Population: Two subjects underwent conditioning regimen
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Bone Marrow and Kidney Transplantation
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Time Frame: 5 years
Description: An adverse event is any occurrence or worsening of an undesirable or unintended sign, symptom, laboratory finding, or disease that occurs during participation in the trial.
  An adverse event will be followed until it resolves or until 30 days after a participant terminates from the study, whichever comes first.
Arm/Group | Combined Bone Marrow and Kidney Transplantation
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Bone Marrow and Kidney Transplantation (N=2)
Thrombotic Microangiopathy (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Bone Marrow and Kidney Transplantation (N=2)
HSV Lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Neutropenia (Immune system disorders) | 1 (1)
Heel pain (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The incidence of adverse events found around 10 days after bone marrow transplant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT02314403/Prot_000.pdf